CLINICAL TRIAL: NCT03104530
Title: Crabmeat and Health Study: Do Brown Crabmeat Consumers Have a Higher Body Burden of Cadmium Compared to Non-crabmeat Consumers?
Brief Title: Crabmeat and Health Study
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: Biomathematics and Statistics Scotland (BioSS) (Unknown); NHS Orkeny (Other)
Responsible Party: Sponsor
Other Study IDs: 2-024-17
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-03

CONDITIONS: Cadmium Body Burden
Keywords: Crab; Brown meat; Cadmium body burden; Ferritin; Zinc; Selenium; Creatinine; B2-Microglobulin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brown crabmeat consumers: Those habitually consuming 40 grams or more of brown crab meat each week.
  Interventions: Other: Brown crabmeat
- Control: Those consuming less than 40 grams of brown crabmeat a year, or no brown crabmeat.

INTERVENTIONS:
Other: Brown crabmeat — Those exposed to higher levels of cadmium due to habitual consumption of 40 grams or more per week of brown meat from crab
  Groups: Brown crabmeat consumers

SUMMARY:
The brown meat from crab may contain high levels of the heavy metal cadmium. Cadmium is found in the environment and long-term exposure can cause accumulation in the body. High cadmium levels can be toxic to the kidney and have been statistically associated with an increased risk of cancer in the lungs, endometrium, bladder, and breast. This study aims to investigate if regular consumers of brown crabmeat have a higher body burden of cadmium than nonconsumers. This is important as no other studies that have addressed this subject. The results of this research may provide guidance on the consumption of brown meat from crab.

The hypothesis of the proposal is that regular habitual consumption of brown crabmeat increases the body burden of cadmium.

This study will recruit 25 healthy participants who consume brown crab meat and 25 healthy participants who do not consume brown crab meat. Volunteers will be eligible if they are ages 40 years and older, non-smokers, and have not had significant occupational exposure to cadmium. Eligibility will be determined using a questionnaire that consenting volunteers will be asked to complete.

Eligible participants will be asked to attend a study visit at the Rowett Institute or at a GP practice in Stromness (depending on participant location). Participants will be weighed and asked to provide a urine sample as well as a 40 ml (2-3 tbsp.) non-fasted blood sample.

The blood and urine samples will be processed at the Rowett Institute or at the Balfour Hospital in Kirkwall (depending on where the study visit took place). Analysis will be completed at the Rowett Institute where whole blood will be analysed for cadmium, selenium, and zinc and the serum for creatinine and ferritin. Urine samples will be measured for cadmium, B2-microglobulin and creatinine.

Recruitment is expected to take place over 4 months. Study participants will have the option of receiving feedback on their cadmium, zinc, selenium and ferritin levels.

DETAILED DESCRIPTION:
Crab meat is low in fat and is a good source of sustainable protein that also provides high levels of minerals (Se, Zn, I), vitamins (B12) and long chain omega-3 fatty acids. However, crab meat can also contain high levels of the heavy metal cadmium (Cd), both in the white meat but especially so in the brown meat (the hepatopancreas and liver). While European legislation sets a limit of 0.5mg Cd/kg wet weight for the white meat from crab, there currently is no limit set for the brown meat from crab due to the large range in concentrations found across member states.

Cd occurs in an inorganic form as an environmental contaminant, both through natural occurrence and from agricultural and industrial sources. The general population is exposed to Cd from various sources, including smoking, but in the non-smoking general population, food is the principal source. Cd is predominantly toxic to the kidney, but it also causes bone demineralisation and is statistically associated with increased risk of cancer in the lung, endometrium, bladder and breast. Moreover, blood Cd levels as low as 0.5 - 0.8 µg/l have been associated with chronic disease. A study of 8,989 US adults from the National Health and Nutrition Examination Survey (NHANES) found such levels to be associated with all-cause mortality, cardiovascular disease, and heart disease after around 5 years follow up and adjustments for a number of potential confounding factors (Tellez-Plaza et al. 2012).

Cd is thought to be absorbed within the body through the use of the same transport pathways as essential metals including zinc, calcium and iron in the intestine. After absorption, Cd is transported in the blood to the liver where it forms a complex with metallothionein, a low molecular weight family of proteins. In the kidney, the Cd-metallothionein complex is filtered in the glomeruli and then reabsorbed in the renal tubules. Although absorption of Cd from the diet in humans is comparatively low (3-5%), it is efficiently retained in the kidney and liver, with a long biological half-life (10 to 30 years). Cd excreted in the urine is a well-characterized exposure biomarker and can be used as a quantitative indicator of cumulative internal dose.

Accumulation of Cd increases with age (Olsson et al, 2002), with 50yrs being the age where urinary cadmium is maximal (WHO/FAO, 2004). Cd is primarily toxic to the kidney, especially to the proximal tubular cells where accumulation over time may cause a decrease in the glomerular filtration rate and eventually, renal failure. Cd causes bone demineralisation, either through direct bone damage or indirectly as a result of renal dysfunction. It is through long term accumulation of Cd that its toxic effects are mainly manifested. As Cd has a high affinity for the main intestinal iron transporter (Kim et al, 2007), the absorption of Cd is influenced by body iron status and there is a close inverse association between serum ferritin (a marker of iron stores) and blood Cd (Berglund et al, 1994). In this regard, studies on human populations have shown increasing blood Cd levels with decreasing serum ferritin in women at fertile age and during pregnancy due to their generally decreased iron status (Berglund et al., 1994).

There is concern that Cd from crab meat consumption can contribute greatly to the body's Cd burden however, no studies have investigated whether the Cd present in crabmeat increases the levels of Cd in the body and similarly, it is not known whether higher Cd intakes in regular crab meat eaters is associated with increased incidence of kidney damage. This study will examine some of these issues. There is evidence from some studies suggesting that selenium and perhaps zinc, which are both present at high levels in crab meat, may counteract the toxicity of Cd (Lindh et al, 1996; Skröder et al, 2015). Moreover, some evidence may suggest that the bioavailability of Cd from crab meat may be less compared to Cd in other foods (Lind et al, 1995). The study will investigate whether volunteers who regularly consume brown crabmeat have higher levels of Cd compared to volunteers who do not consume crabmeat. A frequency questionnaire will be designed to estimate participants' total brown crabmeat intake and to evaluate Cd exposure from crab consumption and this will be compared to the Cd body burden (assessed as urinary Cd and blood Cd levels) to determine whether an association between these variables exists and whether regular crab meat consumers have a higher body burden of Cd compared to non-crabmeat consumers.

HYPOTHESIS

The central hypothesis is that regular habitual consumption of brown crabmeat increases the body burden of cadmium

OBJECTIVES The objective of the study is to determine if regular brown crabmeat consumers have an increased body burden of cadmium compared to non-crabmeat consumers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 40 years and older;
* Regular consumer of brown crab meat (average 40 g per week or greater) or non consumer (> two 60 g portions/year)

Exclusion Criteria:

* Current or ex-smokers in the previous 5 years;
* Those with current or former occupations that result in cadmium exposure (mining, smelter, jewellery or glass making, pain manufacturing, platers/welders, municipal waste incinerators);
* Women who are pregnant;
* Diagnosis of glomerular nephritis or kidney disease;
* Diagnosis of diabetes, hypertension, renal, hepatic, haematological disease, heart/circulation problems, eating disorder or anaemia;
* Vegetarians
* Having given a pint of blood for transfusion purposes within the last month;
* Unsuitable veins for blood sampling;
* Inability to understand the participant information sheet; inability to speak, read and understand the English language.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the public from Aberdeen/Aberdeenshire/Morayshire/Highlands and Orkney.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Cadmium body burden | 1 day of single study visit
  Blood Cd level is a measure of recent Cd intake (2-3 months) and will be measured by closed vessel microwave digestion and inductively coupled plasma mass spectrometry (ICP-MS). Cumulative Cd retention is assessed by measuring Cd in urine (U-Cd) as U-Cd is considered a valid biomarker of lifetime kidney accumulation and will also be measured by ICP-MS.

SECONDARY OUTCOMES:
Zinc status | 1 day of single study visit
  Zinc status will be measured in serum and urine by ICP-MS.
Ferritin | 1 day of single study visit
  Ferritin is a marker of iron stores. Serum ferritin levels will be measured using ELISA as Cd levels (particularly blood-Cd) are known to be inversely related to body iron status and can account for gender differences.
Markers of selenium status | 1 day of single study visit
  Selenium is incorporated into proteins within the body, many of which are antioxidants that protect the body against oxidative damage. Selenium is transported across the body within the protein, selenoprotein P (SEPP-1). Selenium status will be measured by assaying serum selenium levels (by ICP-MS) and by quantification of serum SEPP-1 levels (by an in-house ELISA).
Creatinine | 1 day of single study visit
  Creatinine clearance (calculated using serum and urinary creatinine) is a measure of kidney function. Creatinine in the urine and serum will be analysed using an Assay kit.
B2-microglobulin | 1 day of single study visit
  Urinary levels of B2-microglobulin is a biomarker for kidney toxicity which can be induced by increased body Cd levels. Serum and urine B2-microglobulin will be measured using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Sneddon, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Rowett Institute of Nutrition and Health, Human Nutrition Unit, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No